CLINICAL TRIAL: NCT04767295
Title: PD-1 Monoclonal Antibody Camrelizumab Combined With Albumin Paclitaxel and Platinum for Neoadjuvant Treatment of Adcanced Esophageal Squamous Cell Carcinoma (ESCC): A Single-center, Single-arm Phase II Clinical Study
Brief Title: A Study of Camrelizumab Combined With Chemotherapy as Neoadjuvant Therapy in Adcanced Esophageal Squamous Cell Carcinoma (ESCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-ESCC-001
Record Dates: First submitted 2021-01-18; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: PD-1 Checkpoint Inhibitor; Neoadjuvant Therapy; Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; Carboplatin

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in our study. ESCC participants in this study will be given intravenous administration of SHR-1210 (200mg/3w) combined with albumin paclitaxel (260 mg/m2) plus carboplatin chemotherapy. Every three weeks for a cycle of treatment, which will be conducted twice, and minimally invasive surgery within 5-8 weeks after the last administration. Treatments will be administrated until disease progression, unacceptable adverse events (AE), concomitant diseases that hinder continued treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab, Albumin Paclitaxel, Carboplatin (Experimental): ESCC participants in this study will be given intravenous administration of Camrelizumab (200mg/3w) combined with albumin paclitaxel (260 mg/m2) plus carboplatin chemotherapy. Every three weeks for a cycle of treatment, which will be conducted twice, and minimally invasive surgery within 5-8 weeks after the last administration.
  Treatments will be administrated until disease progression, unacceptable adverse events (AE), concomitant diseases that hinder continued treatment.
  Interventions: Drug: Camrelizumab, Albumin Paclitaxel, Carboplatin

INTERVENTIONS:
Drug: Camrelizumab, Albumin Paclitaxel, Carboplatin — Intravenous administration of Camrelizumab (200mg/3weeks); Intravenous administration of albumin paclitaxel (260 mg/m2/3weeks); Intravenous administration of carboplatin (AUC 4/3weeks)
  Other Names: SHR1210

SUMMARY:
To evaluate the efficacy and safety of camrelizumab combined with albumin paclitaxel and platinum chemotherapy in the preoperative treatment of locally advanced thoracic esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
Primary outcome:

1. Analysis of prognosis efficacy of patients: pathologic complete response (pCR)

Secondary outcome:

Overall survival(OS), Progressive-free survival(PFS), Disease control rate(DCR), Objective response rate(ORR), and the proportion of subjects who completed all treatments and radical resection (R0);

Explorative outcome:

To explore the efficacy of ultrasound gastroscopy, PET/CT, peripheral circulating blood tumor cell (CTC) detection and CTC-based immunofluorescence detection of PD-L1 antibody for the treatment of locally advanced ESCC with camrelizumab combined with albumin paclitaxel and platinum and potential biomarkers for predicting the efficacy of camrelizumab, including but not limited to immunohistochemical detection of PD-L1 expression in tumor specimens, T cell receptor (TCR) sequencing analysis in peripheral blood, and esophageal microbiome Analysis, etc.; patients' quality of life

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before any trial-related procedures are implemented;
* Age 18-70 years, both men and women;
* pathologically confirmed thoracic esophageal squamous cell carcinoma;
* The clinical staging is T3-4a (potentially resectable) N0-2 (PET/CT or cervical, chest and abdomen CT + intra-esophageal ultrasound staging, except those with N3 stage); T1-2N1-2 can be included in the study, T4b, T1-2N0, carcinoma in situ are all excluded;
* The longitudinal length of the tumor is less than 8cm;
* Patients can be followed up for a long time and cooperate with treatment;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; life expectancy> 6 months;
* No other treatments including chemotherapy, radiotherapy, Chinese medicine treatment, etc. were used before selection.
* There is no history of radiotherapy in the chest cavity.
* Hematopoietic function is good before treatment, which is defined as absolute neutrophil count ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90g/L (No blood transfusion within 7 days or no erythropoietin (EPO) dependence);
* Liver function is good before treatment, defined as total bilirubin level ≤ upper normal limit (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 1.5 times ULN;
* Good renal function before treatment, defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); urine protein in routine examination of urine is less than 2+, or 24-hour urine Protein quantitative <1g;
* Good coagulation function before treatment, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, they can also be included in this trail as long as the PT is within the intended range of anticoagulation drugs;
* For female subjects of childbearing age, they should have a negative urine or serum pregnancy test within 3 days before receiving the first study drug administration (cycle 1, day 1). If the urine pregnancy test result cannot be confirmed as negative, blood pregnancy test is required. If there is a risk of conception, male and female patients need to use high-efficiency contraception (ie, a method with a failure rate of less than 1% per year) and continue until at least 180 days after stopping the trial treatment.

Exclusion Criteria:

* Medical history of malignant tumors in other parts, excluding curable non-melanoma skin cancer, radically excised cervical carcinoma in situ, and malignant tumors that have been cured for more than 5 years;
* Pregnant or breast-feeding patients who have fertility but have not taken contraceptive measures;
* Those who are allergic to the study drug camrelizumab, paclitaxel or platinum;
* Previous peripheral neuropathy (whether primary or secondary);
* Severe comorbidities: large-area myocardial infarction, myocardial infarction within 6 months, history of cerebral infarction, heart function ≥ grade III, history of mental illness and severe diabetes, severe pulmonary dysfunction, or other conditions that are not suitable for surgery;
* Participate in other clinical trials at present or within four weeks before being selected;
* Simultaneous treatment with other anti-cancer drugs (including anti-cancer Chinese medicine);
* Have a history of organ transplantation;
* Those who cannot cooperate because of dementia or mental disorders;
* Cachexia, weight loss over the past six months> 10%;
* Histology contains non-squamous carcinoma components, such as small cell carcinoma, adenocarcinoma, etc.;
* Have received the following therapies in the past: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or for another stimulating or synergistic inhibition of T cell receptors (for example, CTLA-4, OX-40, CD137) drug;
* Have received systemic treatment with anti-cancer indications Chinese patent medicines or immunomodulatory drugs (including thymosin, interferon, interleukin) within 2 weeks before the first administration, or received major surgical treatment within 3 weeks before the first administration; those with previous partial gastrectomy, bowel surgery history, or those who are not suitable for minimally invasive surgery are excluded from the group;
* There is clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction; received solid organ or blood system transplantation;
* Active autoimmune diseases that require systemic treatment (such as the use of disease-relieving drugs, corticosteroids, or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
* Diagnosis of immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days before the first administration of the study; physiological dose of glucocorticoids (≤10 mg/ day of prednisone or its equivalent) is allowed;
* Before starting treatment, have not fully recovered from the toxicity and/or complications caused by any intervention (ie ≤ Grade 1 or reach baseline, excluding fatigue or hair loss);
* A history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year before the first administration or current existing in interstitial lung disease;
* Active infections such as tuberculosis that require systemic treatment;
* Known mental illness or drug abuse that may affect compliance with the test requirements;
* Known history of human immunodeficiency virus (HIV) infection (ie HIV 1/2 antibody positive);
* Untreated active hepatitis B; Note: Hepatitis B subjects who meet the following criteria are also eligible for selection: HBV viral load must be <1000 copies/ml (200 IU/ml) before the first dose, and the test Patients should receive anti-HBV therapy during the entire study chemotherapy drug treatment period to avoid viral reactivation. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), prophylactic anti-HBV treatment is not required, but virus reactivation needs to be closely monitored; active Subjects infected with HCV (HCV antibody-positive and HCV-RNA level is higher than the lower limit of detection) ;
* Live vaccine has been vaccinated within 30 days before the first dose (cycle 1, day 1); Note: It is allowed to receive inactivated virus vaccine for seasonal influenza within 30 days before the first administration; however, it is not allowed to receive live attenuated influenza vaccine for intranasal administration;
* The medical history or disease evidence that may interfere with the test results, prevent the subjects from participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator believes are not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | through study completion, an average of 2 year
  evaluated by researchers based on the RECIST 1.1 standard
progression free survival (PFS) | through study completion, an average of 2 year
  evaluated by researchers based on the RECIST 1.1 standard
overall survival (OS) | through study completion, an average of 2 year
  evaluated by researchers based on the RECIST 1.1 standard
Disease control rate(DCR) | through study completion, an average of 2 year
  evaluated by researchers based on the RECIST 1.1 standard
pathologic complete response (pCR) | through study completion, an average of 2 year
  evaluated by researchers based on the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Overall Officials: wangwenxiang@hnca.org.cn wangwenxiang@hnca.org.cn, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Wenxiang Wang, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published work